CLINICAL TRIAL: NCT06223763
Title: An International Retrospective Observational Study Comparing Primary Cytoreductive Surgery With Neoadjuvant Chemotherapy and Interval Cytoreductive Surgery in Patients With Carcinoma of the Ovary, Fallopian Tubes and Peritoneum
Brief Title: SUROVA - Surgery in Ovarian Cancer, Comparing Primary and Interval Cytoreductive Surgery
Acronym: SUROVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Asociación de Amigos de la Universidad de Navarra (Unknown)
Responsible Party: Sponsor
Other Study IDs: SUROVA
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: surgery; gynecology; gynecological surgery; ovarian cancer; neoadjuvant chemotherapy; interval cytoreductive surgery; cytoreductive surgery
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary cytoreductive surgery: Patients underwent primary cytoreductive surgery between January 1, 2018, and December 31, 2019. After that, they underwent adjuvant therapy.
  Interventions: Procedure: Cytoreductive surgery; Drug: Adjuvant chemotherapy
- Interval cytoreductive surgery: Patients underwent primary first course of neoadjuvant chemotherapy between January 1, 2018, and December 31, 2019. After neoadjuvant chemotherapy, the patient underwent interval cytoreductive surgery and then, adjuvant chemotherapy.
  Interventions: Procedure: Cytoreductive surgery; Drug: Neoadjuvant chemotherapy; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Procedure: Cytoreductive surgery — Cytoreductive surgery is a surgical procedure performed with the goal of reducing the tumor burden in the body. This type of surgery is commonly used in the treatment of certain types of cancers, especially in the context of peritoneal carcinomatosis. During cytoreductive surgery, the surgeon attempts to remove as much visible tumor as possible. This may involve the removal of tumors from specific organs and the elimination of tumor lesions on the surface of intra-abdominal organs.
  Other Names: debulking surgery; cytoreduction
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy refers to chemotherapy administered before the primary treatment in cancer management. The goals include reducing tumor size, treating micrometastases, assessing treatment response, converting inoperable tumors to operable ones, and preserving organs or tissues.
  Groups: Interval cytoreductive surgery
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy is chemotherapy given after the primary treatment, such as surgery or radiation therapy, with the aim of eliminating any remaining cancer cells and reducing the risk of recurrence. It is administered to patients who have undergone the initial treatment to enhance the overall effectiveness of the therapy.

SUMMARY:
An international worldwide retrospective cohort observational study comparing primary cytoreductive surgery with neoadjuvant chemotherapy and interval cytoreductive surgery in patients with carcinoma of the ovary, fallopian tubes, and peritoneum.

DETAILED DESCRIPTION:
SUROVA study tries to compare the outcomes of primary cytoreductive surgery with neoadjuvant chemotherapy and interval cytoreductive surgery in patients with carcinoma of the ovary, fallopian tubes, and peritoneum operated between 2018 and 2019 worldwide.

The objective is to know if the surgical approach influences our patients' survival (OS and PFS). To answer this question, SUROVA is necessary.

While the prospective Trust Trial, with results expected in 2024, is designed to address this question, a limitation of this study is that it is confined to patients treated in high-end hospitals. This limitation could introduce bias in the results, as many patients may lack access to such high-level healthcare facilities. Therefore, the objective is to extend the scope of this study to real life. To achieve this, the investigators are seeking to collect data from patients treated globally during 2018 and 2019, involving both primary and interval cytoreduction.

The investigators hope that the results of this study will be subjected to evaluation at international meetings and published in reputable international journals. Authorship will be based on a rigorous criterion tied to the number of valid cases included in the study. Naturally, the aim is to include as many authors as possible.

The researchers strongly believe that patients would greatly benefit from SUROVA data and that it will address this critical question and provide invaluable insights.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 at the time of the surgery.
* Invasive high-grade epithelial ovarian cancer, fallopian tube carcinoma, or primary peritoneal carcinoma in stage International Federation of Gynecology and Obstetrics (FIGO) IIIB-IVB (IVB only if resectable metastases are present), suspected or histologically confirmed and newly diagnosed.
* Patient underwent primary surgery or first course of neoadjuvant chemotherapy between January 1, 2018, and December 31, 2019.
* American Society of Anesthesiologists Physical Status Classification System (ASA) score 1 or 2 at the time of the surgery.
* Surgery performed by laparotomy with an attempt of maximal effort.
* The surgeon must be a certified or non-certified gynecologic oncologist.
* Based on all available information before the surgery (primary or interval), the patient was considered completely resectable.
* Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
* Preoperative imaging (either CT, whole-body MRI, or positron emission tomography (PET)-CT) excluding unresectable disease as per European Society of Gynaecological Oncology (ESGO) criteria.
* Surgical report on residual disease after surgery.

Exclusion Criteria:

* Non-epithelial malignant ovarian neoplasms and borderline tumors.
* Secondary invasive neoplasms in the last 5 years (except synchronal endometrial carcinoma FIGO IA G1/2, non melanoma skin cancer, breast cancer T1 N0 M0 G1/2) or with any signs of relapse or activity.
* Recurrent ovarian cancer.
* Prior chemotherapy for ovarian cancer or abdominal/pelvic radiotherapy.
* Unresectable parenchymal lung metastasis, liver metastasis or bulky lymph-nodes in the mediastinum in CT chest and abdomen/pelvis before surgery (primary or interval).
* Pregnant women at the time of diagnosis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive participant sampling of patients with IIIB-IVB ovarian cancer that underwent primary cytoreductive surgery or interval cytoreductive surgery.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival at 5 years | From date of the first treatment (chemotherapy in the case of neoadjuvant chemotherapy and cytoreduction in the case of primary cytoreductive surgery) to death from ovarian cancer or last follow up, assessed at the 5-year mark.
  Compare overall survival (OS) at 5 years in patients who underwent primary cytoreductive surgery vs. neoadjuvant chemotherapy and interval cytoreductive surgery for stage IIIB-IVB ovarian cancer.

SECONDARY OUTCOMES:
Progression Free Survival at 5 years | From date of the first treatment (chemotherapy in the case of neoadjuvant chemotherapy and cytoreduction in the case of primary cytoreductive surgery) to death from ovarian cancer or last follow up assessed at the 5-year mark.
  Compare Progression Free Survival (PFS) at 5 years in patients who underwent primary cytoreductive surgery vs. neoadjuvant chemotherapy and interval cytoreductive surgery for stage IIIB-IVB ovarian cancer.
Time to first and second subsequent anticancer therapy or death. | From date of the first treatment (chemotherapy in the case of neoadjuvant chemotherapy and cytoreduction in the case of primary cytoreductive surgery) to death from ovarian cancer or last follow up assessed at the 5-year mark.
  Time to first subsequent anticancer therapy is calculated from the date of first treatment (chemotherapy in the case of neoadjuvant chemotherapy and cytoreduction in the case of primary cytoreductive surgery) until the starting date of the first subsequent anticancer therapy or death, whichever occurs first or date of last contact (censored observation). Maintenance treatments following a cytostatic treatment are not considered separate treatment lines.
Information on surgical treatment approaches | Date of last contact up to 5 years
  Gather information on surgical treatment approaches and decision-making processes for patients with advanced high-grade ovarian cancer in worldwide centers
Aletti surgical score | Date of last contact up to 5 years
  Extend the surgery according to the Aletti surgical complexity score, which ranges from 1 to 8, with higher scores indicating more complex surgeries.
Surgical complications: requirement of pharmacological treatment; surgical, endoscopic or radiological intervention, life threatening complications or death. | Date of last contact up to 5 years
  Documentation of surgical complications.
Breast cancer susceptibility gene (BRCA) influence | Date of last contact up to 5 years
  Compare the outcomes between patients with BRCA mutations and those without this mutation
Homologous Recombination Deficiency (HRD) deficiency influence | Date of last contact up to 5 years
  Compare the outcomes between patients with HRD deficiency and those with HRD proficiency

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Chiva, MD, PhD, Study Chair — University of Navarra; Pilar Ordás, PhD student, Study Chair — University of Navarra
Locations (1):
- Clínica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiva L, Ordas P, Martin-Calvo N, Aramendia JM, Sanchez Lorenzo L, Gallego Martinez A, Vizcay A, Minguez JA, Manzour N, Vazquez-Vicente D, Chacon E, Castellanos T, Gonzalez Martin A. An international worldwide retrospective cohort observational study comparing primary cytoreductive surgery with neoadjuvant chemotherapy and interval cytoreductive surgery in patients with carcinoma of the ovary, fallopian tubes, and peritoneum (SUROVA trial). Int J Gynecol Cancer. 2024 Jun 3;34(6):942-945. doi: 10.1136/ijgc-2024-005354. PMID 38479803